CLINICAL TRIAL: NCT03517527
Title: The Effect of The Walking Exercise Training Given According to Transtheoretical Model, and Follow-Up on Improving Exercise Behavior and Metabolic Control in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine KAPLAN SERIN (Other)
Responsible Party: Sponsor-Investigator, Emine KAPLAN SERIN, Assistant Professor, Munzur University
Organization: Munzur University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MunzurU
Record Dates: First submitted 2018-04-09; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Metabolic Control; Walking Exercise; Transtheoretical Model; Nurse
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise
  Other Names: THE WALKING EXERCISE TRAINING GIVEN ACCORDING TO TRANSTHEORETICAL MODEL
  Arms: Intervention

SUMMARY:
OBJECTIVE This study aims to find out the effects of walking exercise training, which is given according to Transtheoretical Model (TTM), and follow-up on improving exercise behavior and metabolic control in type 2 diabetic patients.

RESEARCH DESIGN AND METHODS The study was conducted as a pre-test, post-test experimental model with 76 intervention (INT) groups and 76 control (CON) groups adult type 2 diabetic patients providing the criteria of the study and followed-up by the diabetes polyclinic of Adıyaman Education and Research Hospital. Patient introduction form (PIF), TTM scales and pedometer were used to collect the data. TTM based training was given to the intervention group according to the patients' change stages at hospital 10 weeks once per every 2 weeks. PIF, TTM scales were applied after the training. PIF, TTM scales were applied to the groups 9 months after the pre-test again.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with type-2 diabetes at least six months before, received basic diabetes information, received insulin and/or oral antidiabetic treatment, whose arterial blood pressure was in systolic ≤ 160 mmHg and diastolic ≤ 100 mmHg, who had HbA1c 7% and over, who were literate and had no communication problems were included in the study.

Exclusion Criteria:

* Those who had developed diabetes-related complications (advanced), were pregnant, diagnosed with cancer, had physical and mental problems that prevent walking were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-10-25 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Patient Presentation Form | baseline collected
  The patient presentation form includes questions that question the sociodemographic characteristics and habits of patients, their knowledge of diabetes and its treatment, their exercise status
questions that evaluate the metabolic control variables. | Change from Baseline at 9 months
  FBS, SBS, total cholesterol, HbA1c, LDL, triglyceride, diastolic and systolic BP
Stages of Change for Exercise Questionnaire | Change from Baseline at 9 months
  It was developed by Prochaska and DiClemente, adapted by Marcus et al. to exercise. It was adapted to Turkish society by Ay and Temel in 2007. The scale consists of five questions and reveals the stage of change where the individual in (pre-thinking, thinking, preparation, taking action and maintenance).
Exercise Processes of Change Scale | Change from Baseline at 9 months
  It was developed by Marcus et al. and adapted to Turkish society by Ay and Temel. Exercise Processes of Change Scale is based on a 5-point Likert type and consists of 28 items. The maximum score that an individual can get on the scale is 140, the minimum score is 28. The scale consists of 10 sub-dimensions and 2 main processes (behavioral process and cognitive process) facilitating change involving these sub-dimensions. Cognitive processes are increased awareness, dramatic help, environmental reassessment, self-reassessment, social independence. Behavioral processes are opposition, helping relationships, empowerment management, self-emancipation and stimulus control. The higher scale scores indicate the higher chance of success of the change.
Exercise Self-Efficacy Scale | Change from Baseline at 9 months
  It was developed by Marcus et al. and adapted to Turkish society by Ay and Temel. The scale consists of six items, in the form of five-point Likert. The maximum score that can be taken from the scale is 30 and the minimum score is 6. In the general evaluation of the scale, according to the general average composed of item score averages, the self-efficacy of high-value-average subjects is high, and the self-efficacy of subjects below the average is considered to be low.
Exercise Decisional Balance Scale | Change from Baseline at 9 months
  It was developed by Marcus et al. and adapted to Turkish society by Ay and Temel. There are two sub-dimensions that assess subjective perception including perceived benefits of exercise practice and perceived harmfulness of exercise. The scale is based on 5 point Likert type and consists of 10 items. The overall score of the scale is formed by subtracting the total score of the perceived harmfulness from the total score of the perceived benefit of the exercise practice. The maximum score can be taken from the scale is 20 and the minimum score is -20. The negative result indicates that in the exercise decisional balance, the perceived harmfulness is dominant and the positive result indicates that the perceived benefit of exercise practice is dominant on the scale.